CLINICAL TRIAL: NCT03260608
Title: Randomized Clinical Assessment to Evaluate the Effectiveness of a Psychoeducation and Support Protocol by Telephone, in the Aid of Caregivers of Patients With Dementia in Specialized Ambulatory Accompanying
Brief Title: Effectiveness of a Psychoeducation and Support Protocol by Phone in the Aid of Caregivers of Patients With Dementia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-0326
Record Dates: First submitted 2017-08-16; First posted 2017-08-24 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Dementia
Keywords: dementia, deficits, burden, caregivers, telemedicine.
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: We will select 148 caregivers. Patients will be divided into two groups, both groups will receive printed materials about problematics behaviors in dementia.
  Participants in the intervention group will receive weekly telephone contacts over a period of eight weeks, previously scheduled with psychoeducational and support in the management of their relatives with dementia. Caregivers in the intervention group will have access to a number of phones to spontaneously contact specific guidelines during the eight weeks of intervention.
  Patients from both groups will be interviewed in the baseline, at 8 weeks and 16 weeks.
Who Masked: Outcomes Assessor
Masking Description: The individual who evaluates the outcome(s) of interest in this case the applicators of scales and questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Telesupport: eight weekly phone calls of psychoeducation and support on the illness of their relatives. Patients will also receive printed materials on problematic behaviors about dementia.
  Interventions: Behavioral: Telesupport
- Control (No Intervention): No active intervention. Patients will only receive printed materials on problematic behaviors about dementia and no contact by the research team.

INTERVENTIONS:
Behavioral: Telesupport — In the intervention will be carried out eight weekly phone calls of psychoeducation and support on the disease of the relatives approaching different themes.
  Arms: Intervention

SUMMARY:
Dementias are neurodegenerative syndromes typical of the elderly population and causing a high degree of disability and sick of dependence on others for care. Caregivers of patients with dementia, especially those belonging to the same family suffer with high overhead and is often affected by losses in their own health. The aim of this study is to evaluate the efficacy of a psychoeducation and protocol support, conducted by telephone, in aid of patients with dementia caregivers in specialized outpatient treatment. It will be selected patients in outpatient specialized care. The primary outcome is the change in Zarit Scale.

DETAILED DESCRIPTION:
Dementias are neurodegenerative syndromes typical of the elderly population and cause a high degree of incapacity and dependence of the patient in relation to the care of others. Caregivers of patients with dementia, especially those belonging to the same family, suffer from a high degree of overload, and are often affected by impairments in their own health. Previous studies have shown that telephone interventions for the assistance and guidance of these individuals have a positive impact on their own quality of life as well as on the family members under their care. Measures like this can also optimize specialized services and facilitate the search for medical help when needed.

In this way, the present study aims to evaluate the efficacy of a psychoeducation and support protocol, performed by telephone, to assist caregivers of patients with dementia under specialized outpatient follow-up.

Patients will be divided into two groups. Participants in the intervention group, in addition to the usual primary health care, will receive weekly telephone contacts over a period of eight weeks, previously scheduled with psychoeducational guidelines and support in the management of their relatives and with dementia. The control group will receive the usual follow-up at the in primary health care. Both group will received a prited materials about problematic behavior.

Considering the prevalence and impact of dementia syndromes, it is necessary to conduct studies that are directed at reducing the burden and promoting the information and care of the caregivers of patients with dementia, also providing an improvement in the quality of care. The present project brings as scientific contribution an innovative approach to the reality of our country, with great potential to become an alternative, cost-effective and easily accessible measure for the assistance of people with dementia and their relatives and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* home caregivers
* female and of the same family as the patient
* dementia of any etiology and severity
* caregivers should be responsible for the patient for at least 40 hours per week and for a -minimum period of 6 months
* must have at least 4 years of formal study

Exclusion Criteria:

* caregivers with physical limitations that prevent the application of research instruments
* patients with significant functional impairment related to other diseases
* plans by the caregiver to place the patient in a long-term home in the next 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female caregivers
Enrollment: 148 (Estimated)
Dates: Start 2017-01-15 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the caregiver's level of burden | Week 9
  Zarit Burden Interview
Change from baseline in the caregiver's level of burden | Week 18
  Zarit Burden Interview

SECONDARY OUTCOMES:
Change from baseline in the caregivers's depressive symptoms | Week 9
  Beck Depression Inventory
Change from baseline in the caregivers's depressive symptoms | Week 18
  Beck Depression Inventory
Change from baseline in the caregivers's anxiety symptoms | Week 9
  Beck Anxiety Inventory
Change from baseline in the caregivers's anxiety symptoms | Week 18
  Beck Anxiety Inventory
Change from baseline in the caregivers's quality of life | Week 9
  Quality of Life Questionnaire - WHOQOL
Change from baseline in the caregivers's quality of life | Week 18
  Quality of Life Questionnaire - WHOQOL
Change from baseline in the presence and severity of neurosypsychiatric symptoms in the patient | Week 9
  Neuropsychiatric Inventory - NPI
Change from baseline in the presence and severity of neurosypsychiatric symptoms in the patient | Week 18
  Neuropsychiatric Inventory - NPI
Change from baseline in the patient functionality | Week 9
  Pfeffer Functional Activities Questionnaire
Change from baseline in the patient functionality | Week 18
  Pfeffer Functional Activities Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Artur S Schuh, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: Undecided